CLINICAL TRIAL: NCT01430520
Title: Analgesic Effect of Perioperative Escitalopram for Patients With High Preoperative Level of Pain Catastrophising in Total Knee Arthroplasty
Brief Title: Analgesic Effect of Escitalopram in Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, PHD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THL-04-11; 2011-002034-38 (EudraCT Number); H-3-2011-055 (Registry Identifier: Ethics Committee)
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Tables with Escitalopram (10 mg), 1 tablet a day for 7 days, starting on the day of surgery
  Other Names: Cipralex
  Arms: Escitalopram
Drug: Placebo — Placebo tablets, 1 tablet a day for 7 days, starting on the day of surgery
  Arms: Placebo

SUMMARY:
Pain is a major problem after TKA, especially in patients with high pain catastrophizing. Newer MR-scan studies indicate that Escitalopram may have an immediate cognitive and emotional effect. The investigators therefore investigate the effect of Escitalopram as a perioperative analgesic.

DETAILED DESCRIPTION:
Pain is a major problem after TKA, especially in patients with high pain catastrophizing. Newer MR-scan studies indicate that Escitalopram may have an immediate cognitive and emotional effect. Patients with high pain catastrophizing are mentally vulnerable and may be sensitive to the effects of Escitalopram.

We therefore investigate the effect of Escitalopram as a perioperative analgesic in this group of patients where the pain problem is pronounced.

ELIGIBILITY:
Inclusion Criteria:

* Primary, unilateral total knee arthroplasty (TKA)
* Age > 18 > 81
* Ethnic Danes
* Score > 20 on Pain Catastrophising Scale

Exclusion Criteria:

* Medication that causes risk in combination with SSRI (6 month)
* Treatment for anxiety or depression
* History of depression or mania
* Treatment with systemic glucocorticoids (6 month)
* Treatment with opioids (4 weeks)
* Alcohol or drug abuse
* History of malignancy
* Fertile woman
* History of epilepsia
* Treatment with anticoagulants
* BMI > 40
* Disease affecting central or peripheral nerve function
* Dementia
* History of gastrointestinal bleeding
* History of hepato- or renal insufficiency
* Allergy to Escitalopram

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pain | At 24 hour
  Pain during walking at 24 hour after surgery

SECONDARY OUTCOMES:
Pain | 1 week
  Pain at rest and during walking the first week after TKA
Cumulated pain scores | 1 week
  Cumulated pain scores for pain the first week after TKA
Amount of rescue analgesic | 1 week
  Amount of rescue analgesic the first week after TKA
Side effects | 1 week
  Side effects the first week after TKA
anxiety, depression, and sleep quality | 1 week
  Anxiety, depression, and sleep quality - questionnaire - the first week after TKA
Escitalopram level in blood-sample | 48 hours
  Escitalopram level in blood-sample 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Torben B Hansen, MD, Principal Investigator — Regionshospitalet Holstebro; Henrik Kehlet, MD, Study Director — Rigshospitalet, Denmark; Per W Kristensen, MD, Principal Investigator — Vejle Sygehus; Søren Solgaard, MD, Principal Investigator — Gentofte Hospital; Vibe G Frøkjær, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Gentofte Hospital, Gentofte Municipality, Hellerup
  - Regionshospitalet Holstebro, Holstebro, Holstebro
  - Vejle Sygehus, Vejle, Vejle